CLINICAL TRIAL: NCT04796155
Title: The Use of Intrapartum Ultrasonography in the Evaluation of Labour Arrest in the First and Second Stage
Brief Title: Intrapartum Ultrasonography in Labour Arrest
Acronym: IPUSGLA
Status: Completed | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Arzu Bilge Tekin, Principal Investigator, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Other Study IDs: LAIPUSG
Record Dates: First submitted 2021-03-06; First posted 2021-03-12 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Ultrasonography; Pelvic Floor; Delivery Complication; Maternal-Fetal Relations
Keywords: intrapartum ultrasound; labour arrest; fetal head position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- labour arrest: Pregnant women whose labour progress is delayed and suspected or diagnosed as labour arrest according to the NICE guidelines. Intrapartum ultrasound will be performed at the suspicion of labour arrest in the active phase of the first and second stage of labour. Amniotomy will be performed as routine obstetric care according to the local clinical protocols in accordance with the NICE guideline. Later, diagnosis of labour arrest will be made in slow progress following amniotomy (<1cm cervical dilatation in 2 hours) where a sonographic examination will be repeated.
  Interventions: Diagnostic Test: Intrapartum ultrasound

INTERVENTIONS:
Diagnostic Test: Intrapartum ultrasound — Intrapartum ultrasound will be performed by suprapubic and transperineal approach for 30 seconds.

SUMMARY:
Determination of fetal head position during labour is highly subjective and depends on clinician's experience in vaginal digital examination. Monitoring the progress of labour with intrapartum ultrasound (IU) exhibits higher accuracy rates. However, the dynamic process of labour needs very frequent sonographic examination and that may decrease the feasibility. Consultation to IU at certain time points can positively limit the need for ultrasound, increase the effectiveness of IU and allow for safer labour in consistency with traditional labour management. This study aims to investigate the use of IU in cases with suspected and diagnosed labour arrest in both the first and second stage of labour.

DETAILED DESCRIPTION:
Low-risk pregnant women with singleton, vertex fetus who are at their 36th gestational weeks and above with suspected first and second stages of labour arrest will be enrolled in this study. Intrapartum ultrasound with transperineal and transabdominal approach will be performed at two specific time points; 1) Suspicion of labour arrest, 2) Diagnosis of labour arrest. The fetal head position, station, direction, progression and the structure of pubic arch will be evaluated with IU.

All ultrasound examinations will be monitored and recorded to the memory storage of ultrasound device. Recorded ultrasound examinations will be reviewed and measurements will be performed at the end of the study period by two experienced clinicians who are not involved in the examinations. These two blinded clinicians are not aware of labor outcomes, delivery types, maternal and neonatal outcomes.

General terms are defined according to the NICE guidelines. Those are; the first stage of labour is established when there are regular painful contractions and there is progressive cervical dilatation from 4 cm. If delay in the established first stage is suspected, all aspects of progress in labour are assessed when diagnosing delay, including; cervical dilatation of less than 2 cm in 4 hours for first labours, cervical dilatation of less than 2 cm in 4 hours, or a slowing in the progress of labour for second or subsequent labours, descent, and rotation of the baby's head, changes in the strength, duration and frequency of uterine contractions. Amniotomy is offered to a woman with suspected delay in the established first stage of labour and women are advised to have a vaginal examination 2 hours later, and diagnose delay if progress is less than 1 cm. If oxytocin is used due to insufficient uterine contractions delay is diagnosed as progress is less than 2 cm within 4 hours. With regard to the second stage of labour, for a nulliparous woman; birth would be expected to take place within 3 hours of the start of the active second stage in most women. The delay is diagnosed in the active second stage when it has lasted 2 hours and suspected delay if progress (in terms of rotation and/or descent of the presenting part) is inadequate after 1 hour of the active second stage. For a multiparous woman: birth would be expected to take place within 2 hours of the start of the active second stage in most women. The delay in the active second stage is diagnosed when it has lasted 1 hour for multiparous women and suspected delay if progress (in terms of rotation and/or descent of the presenting part) is inadequate after 30 minutes of the active second stage.

The International Society of Ultrasound in Obstetrics and Gynecology (ISUOG) practical guidelines on intrapartum ultrasound recommend the evaluation of head position and descent during the active phase of labour when labor progress is slow and when operative delivery is considered. The use of IU is not meant to change the classic algorithm of labour monitoring but to provide objective and reliable evaluations of the traditional parameters of crucial importance when prolonged or arrested labour is suspected.

The aim of this study is to evaluate the use of IU in prolonged labour with optimizing the timing of IU.

ELIGIBILITY:
Inclusion Criteria:

* Low-risk pregnant women at their 36th gestational weeks and above
* Singleton, vertex fetus births
* Patients in their active phase of labour in either the first or second phase of labour
* Cases with labour arrest suspicion

Exclusion Criteria:

* Breech presentation
* Multiple pregnancies
* Cases with fetal anomalies
* Intrauterine ex fetus cases
* Patients with vaginismus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women whose active labour progress is prolonged
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Mode of delivery | At the end of delivery
  To predict the mode of delivery; including spontaneous vaginal delivery, operative vaginal delivery, cesarean section

SECONDARY OUTCOMES:
fetal head station | This outcome will be measured twice: (1) During labour after 4 hours of progress if cervical change is 2cm or below. (2) During labour after 2 hours of amniotomy if cervical change is 1cm or below.
  Intrapartum fetal head station will be measured along the longest visible axis of the fetal head, between the intersections with the infrapubic line and the deepest bony part of the fetal head, subtracting 3 cm for the level of the ischial spines.
angle of progression | This outcome will be measured twice: (1) During labour after 4 hours of progress if cervical change is 2cm or below. (2) During labour after 2 hours of amniotomy if cervical change is 1cm or below.
  Angle of progression is defined as the angle existing between a line drawn between the superior and inferior apex of symphysis and a line running from the inferior apex tangentially to the fetal skull contour.
head progression distance | This outcome will be measured twice: (1) During labour after 4 hours of progress if cervical change is 2cm or below. (2) During labour after 2 hours of amniotomy if cervical change is 1cm or below.
  Head progression distance is defined as the longest vertical distance of the fetal cranium from the infrapubic line.
head direction | This outcome will be measured twice: (1) During labour after 4 hours of progress if cervical change is 2cm or below. (2) During labour after 2 hours of amniotomy if cervical change is 1cm or below.
  Head direction is defined as the measurement of the fetal head direction compared to the long axis of the pubic symphysis. Three types of head directions can be determined: ''Head up'', when the line perpendicular to the widest diameter of the head points ventrally at an angle 30, ''Head down'' when this angle is inferior than 0, and ''horizontal'' (all other angles).
rotation angle | This outcome will be measured twice: (1) During labour after 4 hours of progress if cervical change is 2cm or below. (2) During labour after 2 hours of amniotomy if cervical change is 1cm or below.
  Rotation angle will be measured in the transverse plane to identify the midline of the fetal head, defined as the echogenic line interposed between the two cerebral hemispheres. The angle formed by the midline and the anteroposterior diameter of the pubis will be assessed.
occiputospine angle | This outcome will be measured twice: (1) During labour after 4 hours of progress if cervical change is 2cm or below. (2) During labour after 2 hours of amniotomy if cervical change is 1cm or below.
  Occiputospine angle is defined as the degree of fetal head deflection and will be measured by a line tangential to the occipital bone and a line tangential to the first vertebral body of the cervical spine (occiput-spine angle) in a sagittal plane with suprapubic approach.
subpubic arch angle | This outcome will be measured twice: (1) During labour after 4 hours of progress if cervical change is 2cm or below. (2) During labour after 2 hours of amniotomy if cervical change is 1cm or below.
  Subpubic arch angle will be measured between the inferior borders of the pubic rami that converge at the middle of the pubic symphysis.

CONTACTS AND LOCATIONS:
Overall Officials: Murat Yassa, MD, Principal Investigator — Specialist; Niyazi Tug, MD, Study Director — Chief of the department
Locations (1):
- Sehit Prof Dr Ilhan Varank Sancaktepe Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
IPD will be shared upon request after scientific publication

REFERENCES:
- [Background] Blankenship SA, Raghuraman N, Delhi A, Woolfolk CL, Wang Y, Macones GA, Cahill AG. Association of abnormal first stage of labor duration and maternal and neonatal morbidity. Am J Obstet Gynecol. 2020 Sep;223(3):445.e1-445.e15. doi: 10.1016/j.ajog.2020.06.053. PMID 32883453
- [Background] Pergialiotis V, Bellos I, Antsaklis A, Papapanagiotou A, Loutradis D, Daskalakis G. Maternal and neonatal outcomes following a prolonged second stage of labor: A meta-analysis of observational studies. Eur J Obstet Gynecol Reprod Biol. 2020 Sep;252:62-69. doi: 10.1016/j.ejogrb.2020.06.018. Epub 2020 Jun 10. PMID 32570187
- [Background] Ghi T, Eggebo T, Lees C, Kalache K, Rozenberg P, Youssef A, Salomon LJ, Tutschek B. ISUOG Practice Guidelines: intrapartum ultrasound. Ultrasound Obstet Gynecol. 2018 Jul;52(1):128-139. doi: 10.1002/uog.19072. PMID 29974596
- [Background] Bellussi F, Ghi T, Youssef A, Salsi G, Giorgetta F, Parma D, Simonazzi G, Pilu G. The use of intrapartum ultrasound to diagnose malpositions and cephalic malpresentations. Am J Obstet Gynecol. 2017 Dec;217(6):633-641. doi: 10.1016/j.ajog.2017.07.025. Epub 2017 Jul 22. PMID 28743440
- [Background] Dall'Asta A, Angeli L, Masturzo B, Volpe N, Schera GBL, Di Pasquo E, Girlando F, Attini R, Menato G, Frusca T, Ghi T. Prediction of spontaneous vaginal delivery in nulliparous women with a prolonged second stage of labor: the value of intrapartum ultrasound. Am J Obstet Gynecol. 2019 Dec;221(6):642.e1-642.e13. doi: 10.1016/j.ajog.2019.09.045. Epub 2019 Oct 4. PMID 31589867
- See also: NICE guideline — https://www.nice.org.uk/guidance/cg190/resources/intrapartum-care-for-healthy-women-and-babies-pdf-35109866447557